CLINICAL TRIAL: NCT02703766
Title: Pilot Study to Examine the Effects of Weight Gain on Adipose Tissue
Brief Title: Weight Gain and Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-007623
Record Dates: First submitted 2016-01-05; First posted 2016-03-09 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean (Active Comparator): Lean individuals are defined as having body fat content less or equal to 25% in men and less than 35% for women.
  Overfeeding induced weight gain and subsequent weight loss
  Interventions: Behavioral: overfeeding induced weight gain
- Obese (Experimental): obese individuals are defined as having body fat content more than 25% in men and more than 35% for women.
  Overfeeding induced weight gain and subsequent weight loss
  Interventions: Behavioral: overfeeding induced weight gain

INTERVENTIONS:
Behavioral: overfeeding induced weight gain

SUMMARY:
This study aims to examine the role of weight gain in adipose tissue immune cell influx and development of obesity related cardiometabolic disorders. Adipose tissue-mediated chronic systemic inflammation is implicated in the development of cardiometabolic disorders in obesity. Therefore, resolution of adipose tissue inflammation may be key to ameliorating obesity-associated dyslipidemia, insulin-resistance, and cardiovascular disease. Proinflammatory cytokines contribute to the initial influx of immune cells into adipose tissue during weight gain. However, mechanisms regulating these cytokines in the adipose tissue milieu and the effects of weight gain on adipose tissue are not completely understood.

The study proposes to investigate the molecular events contributing to increased infiltration of macrophages and T-cells into adipose tissue during weight gain. The central hypothesis is that in lean subjects (with low body fat mass), healthy fat gain which is associated with decreased expression of proinflammatory cytokines. However, in obesity (high body fat mass), adipose tissue is altered, which permits increased expression of inflammatory cytokines and further fat gain results in influx of immune cells. To test the hypothesis, adipose tissue from well characterized lean (control, with low body fat) and obese individuals (with high body fat) at baseline and after a modest 5% weight gain will be used. Adipose tissue samples after subsequent weight loss will also be examined.

For this study, obesity will be defined by body composition rather than body mass index (BMI), as several studies have shown that BMI does not adequately define obesity and several individuals with normal BMI may indeed have high body fat mass. Individuals with body fat content ≤25% for men, & <35% for women) will be considered lean and individuals with body fat content >25% for men, ≥35% for women will be considered obese.

ELIGIBILITY:
Inclusion Criteria

* Age: 18 to 40 (inclusive) years
* BMI 18.5 <30 kg/m2
* Gender: Both males and females will be allowed to participate in the study
* Predominantly sedentary
* Absence of any chronic medical conditions other than seasonal or environmental allergies
* On no prescription medications other than second generation antihistamines (cetirizine , Fexofenadine, Desloratadine, Loratadine, etc), oral contraceptive pills, or intrauterine devices
* Not a current smoker or tobacco user
* Not pregnant or breast feeding and not intending to become pregnant or breast feed
* Lean (low body fat mass) (body fat content ≤ 25% for men, < 35% for women) n=7; Obese (high body fat mass) (body fat content >25% for men, ≥ 35% for women) n=7
* Ability to provide written informed consent

Exclusion Criteria

* Vulnerable study population will be excluded
* Presence of chronic diseases such as diabetes, and cardiovascular disease
* Pregnancy
* Anemic (hemoglobin <13.5 g/dL for men and <12.0 g/dL for women)
* Postmenopausal
* Smoking
* Use of chronic Medications (aspirin, statin, anti-inflammatory drugs)
* Subjects found to have significant sleep disorders will be excluded
* Dietary restrictions including lactose intolerance, and vegan diet
* Eating disorders that may interfere with weight gain and weight loss

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in adipose tissue inflammation by 8 week of modest weight gain followed by 8 week of weight loss. | 16-20 weeks
  Adipose tissue inflammation will be measures by RTPCR and Western Blot. These will be presented as ratio to endogenous house keeping gene.

SECONDARY OUTCOMES:
Change from baseline in blood pressure by 8 week of modest weight gain followed by 8 weeks of weight loss. | 16-20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided